CLINICAL TRIAL: NCT03849066
Title: Enhancing Medication Safety in Children With Polypharmacy Using Parent- Reported Symptom Assessments
Brief Title: Parent-Reported Symptom Assessments in Children Taking Multiple Medications
Acronym: PRSA
Status: Completed | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Other Study IDs: 16-2538; 5K23HD091295 (NIH)
Record Dates: First submitted 2019-02-14; First posted 2019-02-21 (Actual); Results first posted 2023-02-21 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-01

CONDITIONS: Neurologic Disorder; Chronic Disease; Pediatric Disorder
Keywords: Neurological Impairment; Pediatric Complex Chronic Condition; Children with Medical Complexity; Pediatric Polypharmacy
MeSH Terms: conditions — Nervous System Diseases; Chronic Disease; Neurologic Manifestations

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cross-Sectional PRSA: This will be a cross-sectional analysis of children with neurological impairment and polypharmacy.
  Interventions: Other: Parent-Reported Symptom Assessment

INTERVENTIONS:
Other: Parent-Reported Symptom Assessment — As the basis for PRSA, the investigator will use the PediQuest Memorial Symptom Assessment Scale (PQ-MSAS), which is an adapted pediatric-specific version of the validated adult MSAS that assesses 28 physical and psychological symptoms over the past week. The study instrument is designed to be completed by a full-proxy parent, and 2 versions tailored for specific age groups are available (0-3, 3-18 years-old). Spanish versions are available for both instruments. The PQ-MSAS contains 28 symptom items, each with 4-point scores for domains of frequency, severity, and extent of bother. Based on these components, a global symptom score and individual symptom scores can be calculated (0-100 scale, with 100 being the worst).
  Other Names: PRSA

SUMMARY:
This study plans to learn about how to measure symptoms (like tiredness or rash) in children with special healthcare needs who take 5 or more medications. Sometimes symptoms change in severity over time or new symptoms develop. This can happen after a new medication is started. This can also happen after the dose of an existing medication is changed. The Investigators believe that parents will be able to provide the best assessment of any symptoms that their child might be experiencing. This study asks parents to report any symptoms their child is currently experiencing.

DETAILED DESCRIPTION:
An increasing number of children with complex chronic conditions (CCCs) who have intractable illnesses or multi-organ dysfunction are exposed to daily polypharmacy. Parents of children with polypharmacy often administer 5 or more medications each day, sometimes for months, including high-risk medications prescribed by many different specialists in multiple settings of care. While medications can be life-saving, polypharmacy increases the risk of additive adverse effects, drug-drug interactions, and can lead to serious adverse drug events (ADEs). Pediatric ADEs result in over 4.3 million estimated ambulatory visits annually, including >150,000 pediatric emergency room visits. Despite the risks associated with polypharmacy, little is known about how polypharmacy escalates and how polypharmacy should be managed. To enable children to thrive at home using medications while minimizing unwanted symptoms, this proposal aims to implement a prospective, parent-reported symptom assessment system to guide and monitor pharmaceutical care for high-risk children. Strategies to improve recognition of problematic symptoms will have a substantial impact on the health of children.

ELIGIBILITY:
Inclusion Criteria:

* Neurological impairment
* 5 or more scheduled medications
* English- or Spanish-speaking

Exclusion Criteria:

* Receives primary care outside outside of the Children's Hospital Colorado Network of Care

Ages: 1 Day to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: All patients with neurological impairment and 5 or more scheduled medications aged 0-17 years-old (inclusive) and their parents will be included.
Sampling Method: Non-Probability Sample
Enrollment: 136 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2022-08-01 (Actual); Study Completion 2022-08-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James A Feinstein, MD MPH, Principal Investigator — Associate Professor of Pediatrics
Locations (1):
- Children's Hospital Colorado, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No
Any and all data collected as part of this project will be released in accordance with standard data sharing policies and procedures. All data will be made available in a timely manner to the broader scientific community after study results are published as manuscripts in peer-reviewed journals. All data released will be de-identified, with no information that could be linked to any participating patients or caregivers in order to ensure the confidentiality of all study participants.
  The main deliverable of this research will be a parent-reported system assessment system tailored to the needs of children with polypharmacy that will be ready for definitive evaluation. After the results from this study are published, upon request, the investigator will readily and willingly make available any and all data management tools, study instruments, and analytic programs used in the project.

REFERENCES:
- [Background] Feinstein JA, Feudtner C, Valuck RJ, Kempe A. The depth, duration, and degree of outpatient pediatric polypharmacy in Colorado fee-for-service Medicaid patients. Pharmacoepidemiol Drug Saf. 2015 Oct;24(10):1049-57. doi: 10.1002/pds.3843. Epub 2015 Aug 7. PMID 26248529
- [Background] Feinstein J, Dai D, Zhong W, Freedman J, Feudtner C. Potential drug-drug interactions in infant, child, and adolescent patients in children's hospitals. Pediatrics. 2015 Jan;135(1):e99-108. doi: 10.1542/peds.2014-2015. Epub 2014 Dec 15. PMID 25511114
- [Background] Feinstein JA, Feudtner C, Kempe A. Adverse drug event-related emergency department visits associated with complex chronic conditions. Pediatrics. 2014 Jun;133(6):e1575-85. doi: 10.1542/peds.2013-3060. Epub 2014 May 19. PMID 24843054
- [Background] Berry JG, Poduri A, Bonkowsky JL, Zhou J, Graham DA, Welch C, Putney H, Srivastava R. Trends in resource utilization by children with neurological impairment in the United States inpatient health care system: a repeat cross-sectional study. PLoS Med. 2012 Jan;9(1):e1001158. doi: 10.1371/journal.pmed.1001158. Epub 2012 Jan 17. PMID 22272190
- [Background] Dussel V, Orellana L, Soto N, Chen K, Ullrich C, Kang TI, Geyer JR, Feudtner C, Wolfe J. Feasibility of Conducting a Palliative Care Randomized Controlled Trial in Children With Advanced Cancer: Assessment of the PediQUEST Study. J Pain Symptom Manage. 2015 Jun;49(6):1059-69. doi: 10.1016/j.jpainsymman.2014.12.010. Epub 2015 Jan 30. PMID 25640275
- [Background] Wolfe J, Orellana L, Cook EF, Ullrich C, Kang T, Geyer JR, Feudtner C, Weeks JC, Dussel V. Improving the care of children with advanced cancer by using an electronic patient-reported feedback intervention: results from the PediQUEST randomized controlled trial. J Clin Oncol. 2014 Apr 10;32(11):1119-26. doi: 10.1200/JCO.2013.51.5981. Epub 2014 Mar 10. PMID 24616307
- [Background] Feinstein JA, Morrato EH, Feudtner C. Prioritizing Pediatric Drug Research Using Population-Level Health Data. JAMA Pediatr. 2017 Jan 1;171(1):7-8. doi: 10.1001/jamapediatrics.2016.3462. No abstract available. PMID 27893067
- [Result] Feinstein JA, Feudtner C, Kempe A, Orth LE. Anticholinergic Medications and Parent-Reported Anticholinergic Symptoms in Neurologically Impaired Children. J Pain Symptom Manage. 2023 Feb;65(2):e109-e114. doi: 10.1016/j.jpainsymman.2022.10.013. Epub 2022 Nov 2. PMID 36332769
- [Result] Marquez C, Thompson R, Feinstein JA, Orth LE. Identifying opportunities for pediatric medication therapy management in children with medical complexity. J Am Pharm Assoc (2003). 2022 Sep-Oct;62(5):1587-1595.e3. doi: 10.1016/j.japh.2022.04.005. Epub 2022 Apr 12. PMID 35527209
- [Result] Feinstein JA, Friedman H, Orth LE, Feudtner C, Kempe A, Samay S, Blackmer AB. Complexity of Medication Regimens for Children With Neurological Impairment. JAMA Netw Open. 2021 Aug 2;4(8):e2122818. doi: 10.1001/jamanetworkopen.2021.22818. PMID 34436607
- [Result] Feinstein JA, Feudtner C, Blackmer AB, Valuck RJ, Fairclough DL, Holstein J, Gregoire L, Samay S, Kempe A. Parent-Reported Symptoms and Medications Used Among Children With Severe Neurological Impairment. JAMA Netw Open. 2020 Dec 1;3(12):e2029082. doi: 10.1001/jamanetworkopen.2020.29082. PMID 33306117
- [Result] Feinstein JA, Feudtner C, Valuck RJ, Fairclough DL, Holstein JA, Samay S, Kempe A. Identifying Important Clinical Symptoms in Children With Severe Neurological Impairment Using Parent-Reported Outcomes of Symptoms. JAMA Pediatr. 2020 Nov 1;174(11):1114-1117. doi: 10.1001/jamapediatrics.2020.2987. PMID 33044500
- [Result] Feinstein JA, Orth LE. Making Polypharmacy Safer for Children with Medical Complexity. J Pediatr. 2023 Mar;254:4-10. doi: 10.1016/j.jpeds.2022.10.012. Epub 2022 Oct 15. PMID 36252865

RESULTS

PARTICIPANT FLOW:
Recruitment Details: We obtained parental written informed consent and enrolled and assessed English-speaking and Spanish-speaking children aged 0 to 17 years with SNI and polypharmacy (≥5 medications) who received primary care in a large, hospital-based special health care needs clinic.
Groups:
- Parent Reported Symptom Assessment (PRSA): This is a cross-sectional analysis of children with neurological impairment and polypharmacy. As the basis for PRSA, the investigator will use the PediQuest Memorial Symptom Assessment Scale (PQ-MSAS), which is an adapted pediatric-specific version of the validated adult MSAS that assesses 28 physical and psychological symptoms over the past week. The study instrument is designed to be completed by a full-proxy parent, and 2 versions tailored for specific age groups are available (0-3, 3-18 years-old). Spanish versions are available for both instruments. The PQ-MSAS contains 28 symptom items, each with 4-point scores for domains of frequency, severity, and extent of bother. Based on these components, a global symptom score and individual symptom scores can be calculated (0-100 scale, with 100 being the worst).
Period: Overall Study
Arm/Group | Parent Reported Symptom Assessment (PRSA)
Started | 136
Completed | 123
Not Completed | 13

BASELINE CHARACTERISTICS:
Population: 13 participants enrolled but did not complete the study activities and were excluded from analysis.
Arm/Group | Parent Reported Symptom Assessment (PRSA)
Number analyzed (Participants) | 123
Age, Continuous [Median (Inter-Quartile Range); unit: years] — Population: 13 participants enrolled but did not complete the study activities and were excluded from analysis.
  years | 9 [5 to 12]
Sex: Female, Male [Count of Participants; unit: Participants] — Population: 13 participants enrolled but did not complete the study activities and were excluded from analysis.
  Participants
    Female | 50
    Male | 73
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: 13 participants enrolled but did not complete the study activities and were excluded from analysis.
  Participants
    Hispanic or Latino | 29
    Not Hispanic or Latino | 94
    Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: 13 participants enrolled but did not complete the study activities and were excluded from analysis.
  Participants
    American Indian or Alaska Native | 1
    Asian | 0
    Native Hawaiian or Other Pacific Islander | 0
    Black or African American | 5
    White | 94
    More than one race | 17
    Unknown or Not Reported | 6
Region of Enrollment [Number; unit: participants] — Population: 13 participants enrolled but did not complete the study activities and were excluded from analysis.
  participants
    United States | 123
Complex Chronic Condition (CCC) Count [Count of Participants; unit: Participants] — Population: 13 participants enrolled but did not complete the study activities and were excluded from analysis.
  Participants
    1-2 | 49
    3-4 | 55
    5 or More | 19

OUTCOME MEASURES:

1. Primary Outcome: Global Symptom Score
Description: As the basis for PRSA, we used the PediQuest Memorial Symptom Assessment Scale (PQ-MSAS), which is an adapted pediatric-specific version of the validated adult MSAS that assesses 28 physical and psychological symptoms over the past week. The study instrument is designed to be completed by a full-proxy parent, and 2 versions tailored for specific age groups are available (0-3, 3-18 years-old). Spanish versions are available for both instruments. The PQ-MSAS contains 28 symptom items, each with 4-point scores for domains of frequency, severity, and extent of bother. Based on these components, a global symptom score and individual symptom scores can be calculated (0-100 scale, with 100 being the worst).
Time Frame: Baseline
Population: We obtained parental written informed consent and enrolled and assessed English-speaking and Spanish-speaking children 0-17 years-old (inclusive) with SNI and polypharmacy (≥5 medications) who received primary care in a large, hospital-based special health care needs clinic.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Parent Reported Symptom Assessment (PRSA)
Number analyzed (Participants) | 123
score on a scale | 12.1 [5.4 to 20.8]

2. Secondary Outcome: Medication Count
Description: Prescription and over-the-counter medications were counted at the time of the visit. To reflect parent-facing medication complexity, we excluded clinic-administered or inpatient-administered medications (eg, vaccines or botulinum toxin injections).
Time Frame: Baseline
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Parent Reported Symptom Assessment (PRSA)
Number analyzed (Participants) | 123
Participants
  5-9 Medications | 25
  10-14 Medications | 44
  15 or More Medications | 54

3. Secondary Outcome: Medication Regimen Complexity Index Score (MRCI)
Description: MRCI scores were calculated automatically from EHR data using the MRCI tool, scoring instructions, and examples that are publicly available. Conceptually, the total MRCI score for a CMR is the sum of 3 weighted subscores (dosage form, dose frequency, and specialized instructions), with increasing weights corresponding to the difficulty of administration. The minimum total MRCI score for a participant using a single medication is 1.5. The total MRCI score has no upper limit because it is dependent on the total number of medications, and higher MRCI scores indicate more-complex regimens.
Time Frame: Baseline
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Parent Reported Symptom Assessment (PRSA)
Number analyzed (Participants) | 123
score on a scale | 46 [8 to 139]

ADVERSE EVENTS:
Time Frame: This was a cross-sectional analysis and adverse events were not monitored/assessed longitudinally after completion of the study visit.
Description: All-Cause Mortality, Serious, and Other (Not Including Serious) Adverse Events were not monitored/assessed.
Arm/Group | Parent Reported Symptom Assessment (PRSA)
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

LIMITATIONS AND CAVEATS:
13 participants enrolled but did not complete the study activities and were excluded from analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-01-07): https://cdn.clinicaltrials.gov/large-docs/66/NCT03849066/Prot_SAP_000.pdf